CLINICAL TRIAL: NCT06521372
Title: NiOS (Non-Invasive Oocyte Sorting) Study
Brief Title: The Aim of This Study is to Determine if Oocyte Sorting for Group Culture Using an Artificial Intelligence Image Analysis Tool (MagentaTM) Increases the Usable Blastocyst Yield and Subsequent Pregnancy in Patients Undergoing IVF
Acronym: NiOS
Status: Recruiting | Type: Observational
Sponsor: Ovation Fertility (Other)
Collaborators: Future Fertility Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OVA-11-2023-TX
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Infertility Primary
Keywords: Artificial Intelligence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oocytes with AI: Oocytes assessed by the Magenta software
  Interventions: Other: Magenta AI image analysis tool
- Oocytes without AI: Oocytes randomly selected

INTERVENTIONS:
Other: Magenta AI image analysis tool — MagentaTM is a non-invasive image analysis tool that utilizes artificial intelligence to evaluate 2-dimensional images of denuded mature MII oocytes. The MagentaTM software has been analyzed retrospectively, by Future Fertility. This data displays that a higher MagentaTM score is associated with a higher chance of blastocyst development. Additionally, the MagentaTM software has been validated in a prospective multi-center study, displaying that a higher MagentaTM score correlates to a higher chance of blastocyst development.
  Groups: Oocytes with AI

SUMMARY:
The aim of this study is to determine if oocyte sorting for group culture using an artificial intelligence image analysis tool (MagentaTM) increases the usable blastocyst yield and subsequent pregnancy in patients undergoing IVF.

DETAILED DESCRIPTION:
Introduction Magenta™ is a software image analysis tool developed by Future Fertility that allows personalized reproductive prediction for each oocyte (egg cell) analyzed. It is a cloud-based software that was developed to assess the probability of an oocyte to fertilize and develop into a blastocyst (ball of rapidly dividing cells that will become an embryo). It is a non-invasive image analysis tool that uses artificial intelligence (AI) to predict outcomes based on a single 2-D image of a mature oocyte (denuded oocyte) prior to freezing or sperm injection (ICSI). Magenta™ was designed and built specifically to analyze oocytes in the IVF lab. It was created based on more than 20,000 images of oocytes and their known reproductive outcomes. It is an image analysis neural network that can identify important signals beyond the limited morphological features detected by embryologists, like facial recognition systems in use today. Without the development of this AI tool, there are no standard assessments for oocyte quality within the IVF process. The use of Magenta™ in this study is investigational.

In standard IVF laboratories, oocytes can undergo their developmental period alone (single culture) or be grouped with other oocytes during this time (group culture). Research has shown that group culture has some developmental advantages over single culture.

What is this study for? At the moment, there is no standard method to sort oocytes into groups for their developmental period. Currently, oocytes are sorted in a random manner. We hope that Magenta™ analysis will provide information at this early stage of development and inform a better way to sort oocytes into groups (from lowest to highest quality). The objective of this research study is to compare sorting the oocytes randomly to utilizing the MagentaTM tool for oocyte assessment to determine which oocytes should be grouped together. Study participants will be randomly assigned to the control (random sorting) or the study (Magenta™ analysis) groups at the time of oocyte retrieval. You have an equal chance of being assigned to either group. We intend to enroll 450 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Fresh MII oocytes
* ICSI cycles with patient's or donor's sperm
* Patient's or donor's oocytes
* Full IVF cycle information available (including total number of oocytes retrieved, total MII oocytes, fertilization, embryo and blastocyst development, as well as ploidy status or implantation results, and 6-7 week ultrasound, if applicable)
* Good quality images of MII oocytes taken with a specified camera (Basler) and Future Fertility Software
* Single embryo transfers (SETs) at blastocyst stage.
* Blastocyst freeze-all cycles

Exclusion Criteria:

* Severe male factor infertility (<1 million motile), including surgically retrieved sperm.
* ICSI cycles inseminating in vitro matured (IVM) oocytes
* Rescue ICSI oocytes (oocytes failed standard IVF and are re-inseminated by ICSI)
* Low quality images - Poor quality images on day of upload or before unblinding
* Lack of correlating reproductive outcomes (full IVF lab results not available).
* Autologous or donor frozen/warmed oocytes
* Day 3 embryo transfers or cleavage stage embryo freezing
* Patients with less than 6 mature oocytes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients seeking IVF treatment
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Compare blastocyst development rate | 5 to 7 days
  Blast Development rates between oocytes (and resulting embryos) that are group cultured according to MagentaTM scores versus oocytes (and resulting embryos group) cultured as per the standard of care following random sorting. Blastocyst development is defined by an embryologist's grading, according to the laboratory's grading system.

SECONDARY OUTCOMES:
Fertilization Rate | 1Day
  within each MagentaTM score group and random sorting groups.
Morphological Blastocyst Quality | 7 days
  within each MagentaTM score group and random sorting groups.
Euploidy Rate | 14 days
  within each MagentaTM score group and random sorting groups.
Pregnancy Rate | 6 weeks
  Positive pregnancy test

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ovation Fertility Las Vegas, Las Vegas, Nevada
  - Ovation Fertility Cincinnati, Cincinnati, Ohio
  - Ovation Fertility - Nashville, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided
Pending results